CLINICAL TRIAL: NCT00871078
Title: Anatomic and Visual Function Assessments on Asymptomatic HIV-positive Patients Using Optical Coherence Tomography and Frequency Doubling Technology Perimetry
Brief Title: Anatomic and Visual Function Assessments on Asymptomatic HIV-positive Patients
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Tiago Eugênio Faria e Arantes, Federal University of São Paulo
Other Study IDs: BRA-713/06
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: HIV-positive patients with CD4 cell counts below 100 cells/mm³ at some point of time in their medical history lasting for at least 6 months
  Interventions: Device: Optical Coherence Tomography (OCT); Device: Frequency Doubling Technology (FDT) perimeter
- B: HIV-positive patients with CD4 cell counts never below 100 cells/mm³ in their medical records
  Interventions: Device: Optical Coherence Tomography (OCT); Device: Frequency Doubling Technology (FDT) perimeter
- C: HIV-negative patients (control group)
  Interventions: Device: Optical Coherence Tomography (OCT); Device: Frequency Doubling Technology (FDT) perimeter

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — Macular and retinal nerve fiber layer OCT (Stratus OCT, Carl Zeiss Meditec, Dublin, CA) will be performed both in patients and controls
Device: Frequency Doubling Technology (FDT) perimeter — 24-2 FDT Threshold (Humphrey Matrix, Carl Zeiss Meditec, Dublin CA; Welch-Allyn, Skaneateles, NY) will be performed both in patients and controls.

SUMMARY:
The purpose of this study is to assess retinal nerve fiber layer thickness and macular thickness measured with optical coherence tomography (OCT) on patients infected by HIV virus without ocular manifestations and to correlate these results with perimetric findings assessed by frequency doubling technology perimetry (FDT).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AIDS
* Best-corrected visual acuity 20/25 or better
* Refractive error of 0±5.0 diopters and astigmatism of 0±3.0 diopters
* Normal intraocular pressure (≤21mmHg)

Exclusion Criteria:

* Cataract or any visible media opacity
* HIV-related infectious retinopathy
* Risk factors for the development of glaucoma

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV infected patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Arantes, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo (UNIFESP/EPM), São Paulo, São Paulo, Brazil